CLINICAL TRIAL: NCT07184125
Title: Effect of Midazolam as Premedication in Patients Undergoing Breast Conservation Study
Status: Completed | Type: Observational
Sponsor: Shaukat Khanum Memorial Cancer Hospital & Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-23-27
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2024-08

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 01 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1 group will be given Midazolam: 2nd group will be given normal saline
  Interventions: Drug: To measure anxiolysis, satisfaction level of patient after receiving Midazolam

INTERVENTIONS:
Drug: To measure anxiolysis, satisfaction level of patient after receiving Midazolam — Anxiety & satisfaction

SUMMARY:
Patient are randomized into 2 groups under computer registered numbers. Patient anxiety score is calculated through APAIS SCORE. Then one group is given Midazolam, and the other group is given normal saline and then after one day patients satisfaction is calculated through Lppsq scale.

DETAILED DESCRIPTION:
Patient are randomized into 2 groups under computer registered numbers. After taking approval from hospital ethical committee, 124 females fulfilling inclusion criteria are selected. All patients will receive written information about the study on the day before surgery and before signing informed consent. Patient anxiety score is calculated through APAIS SCORE. Then one group is given Midazolam, and the other group is given normal saline and then after one day patients satisfaction is calculated through Lppsq scale.

ELIGIBILITY:
Inclusion Criteria:

1. All patients undergoing breast conservation surgery
2. ASA I-II

Exclusion Criteria:

1. Patients already on anxiolytic medication
2. Pregnancy
3. Allergy to Midazolam,
4. Patient with diagnosed psychosis,
5. Chronic kidney disease.

Max Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 124
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Comparison of frequency of patient satisfaction & anxiety | 1 day
  It is a single blinded randomized control trial 124 adult females scheduled for surgery, were randomized to receive either Intravenous Midazolam or single Placebo before anesthesia induction. Pre and post medication anxiety levels on day of surgery will be assessed on APAIS score. Post operative satisfaction will be assessed on first post operative day using Lppsq.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mehwish Shafique, MBBS, FCPS Anesthesia, Principal Investigator — Shaukat Khanam Cancer Memorial Hospital & Research Centre
Locations (1):
- Shaukat Khanam Cancer Memorial Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Dr. Ahsun Waqar, Dr. Saad Ur Rehman, Dr. Huma Saleem
Supporting Information: ICF
Time Frame: Till the end of study
Access Criteria: All investigators, to help in analyzing the data.